CLINICAL TRIAL: NCT05876065
Title: Efficacy and Safety of Capecitabine and Cyclophosphamide (XC) Versus Physician's Choice as Maintenance Therapy for Advanced Breast Cancer: a Randomized, Controlled, Open-label Clinical Trial
Brief Title: Capecitabine and Cyclophosphamide (XC) as Maintenance Therapy for Advanced Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wenjin Yin (Other)
Responsible Party: Sponsor-Investigator, Wenjin Yin, Deputy Chief of Breast Surgery Department, RenJi Hospital
Organization: RenJi Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY2023-073-A
Record Dates: First submitted 2023-05-14; First posted 2023-05-25 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- capecitabine and cyclophosphamide (XC) (Experimental): capecitabine and cyclophosphamide as maintenance therapy every 3 weeks
  Interventions: Drug: XC
- physician's choice (Active Comparator): Any physician's choice as maintenance therapy (except for XC regimen).
  Interventions: Drug: TPC

INTERVENTIONS:
Drug: XC — Capecitabine (bid po, d1-14) and cyclophosphamide (qd po, d1-d14) every 21 days
  Arms: capecitabine and cyclophosphamide (XC)
Drug: TPC — Any physician's choice as maintenance therapy (except for XC regimen)
  Arms: physician's choice

SUMMARY:
To compare the efficacy and safety of capecitabine and cyclophosphamide (XC) versus physician's choice as maintenance therapy for patients with advanced breast cancer who achieved disease control after salvage treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female, age≥18 years old
* ECOG≤2
* Pathologically confirmed primary breast cancer, with pathologically or radiologically confirmed recurrent or metastatic lesions
* HR+/HER2+ or HR-/HER2+ or HR-/HER2-
* At least one measurable lesion or bone-only disease (osteolytic or mixed) according to RECIST v1.1
* Disease control (complete response + partial response + stable disease) after salvage treatment
* Expected survival ≥6 months
* Adequate organ function

Exclusion Criteria:

* during pregnancy and lactation
* Patients with central nervous system metastasis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From the date of starting maintenance therapy to the date of first documentation of disease progression or death from any cause (up to approximately 1 year)
  PFS is defined as the time from the date of starting maintenance therapy to the date of disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Adverse events | From the date of starting maintenance therapy to the end of the treatment (up to approximately 1 year)]
  Adverse events during maintenance therapy will be assessed according to the NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Wenjin Yin, M.D., Principal Investigator — Renji Hospital,School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No